CLINICAL TRIAL: NCT01277016
Title: A Randomized Open-label Multicenter Phase III Trial of Melphalan and Dexamethasone (MDex) Versus Bortezomib, Melphalan and Dexamethasone (BMDex) for Untreated Patients With Systemic Light-chain (AL) Amyloidosis
Brief Title: A Trial for Systemic Light-chain (AL) Amyloidosis
Acronym: EMN-03
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Myeloma Network B.V. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMN-03; 2010-022395-31 (EudraCT Number)
Record Dates: First submitted 2011-01-10; First posted 2011-01-14 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2016-08

CONDITIONS: AL Amyloidosis
Keywords: Amyloidosis; Bortezomib
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Amyloidosis | interventions — Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MDex: (No Intervention): MDex:
  Administration of oral melphalan (M) at 0.22 mg/kg and dexamethasone (Dex) at 40 mg daily for 4 consecutive days every 28 days (MDex) until end of therapy
- BMDex (Experimental): BMDex:
  cycles 1 and 2 = MDex with bortezomib (B) at 1.3 mg/m2 i.v. on days 1, 4, 8 and 11 of a 28 day cycle, cycles 3 - 8 = MDex with bortezomib at 1.3 mg/m2 i.v. on days 1, 8, 15 and 22 of a 35 day cycle.
  Interventions: Drug: BMDex

INTERVENTIONS:
Drug: BMDex — BMDex:
  cycles 1 and 2 = MDex with bortezomib (B) at 1.3 mg/m2 i.v. on days 1, 4, 8 and 11 of a 28 day cycle, cycles 3 - 8 = MDex with bortezomib at 1.3 mg/m2 i.v. on days 1, 8, 15 and 22 of a 35 day cycle.
  Other Names: Bortezomid; Melphalan; Dexametasone
  Arms: BMDex

SUMMARY:
In this multi-center phase III trial, untreated patients diagnosed with AL who are not candidates for stem cell transplant with melphalan 200 mg/m2 are the target population. Stage I and II patients will be eligible. Stage III patients will be enrolled in an ancillary phase II study. Eligible patients will be stratified as cardiac stage I or stage II and then randomized to receive MDex or BMDex.

Primary objective is to compare hematologic(clonal) response i.e. the rate of complete response (CR) + partial response (PR) defined according to the criteria of the International Society for Amyloidosis consensus.

DETAILED DESCRIPTION:
Design In this multi-center phase III trial, untreated patients diagnosed with AL who are not candidates for stem cell transplant with melphalan 200 mg/m2 are the target population. Patients who are eligible for SCT with melphalan 200 mg/m2 but who decline to undergo transplantation will be enrolled in the study as a subgroup with stratified randomization. Because many newly diagnosed AL patients present with limited organ reserve, the eligibility criteria take into consideration the impact of cardiac involvement on overall survival using cardiac biomarker staging. Stage I and II patients will be eligible. Stage III patients will be enrolled in an ancillary phase II study. Eligible patients will be stratified as cardiac stage I or stage II and then randomized to receive MDex or BMDex.

Intervention Untreated patients with AL amyloidosis will be offered treatment on this study. After being screened and found eligible, patients will be stratified based on cardiac stage as stage I or stage II. Thresholds for cTnT, cTnI, and NT-proBNP are <0.035 microg/L, <0.1 microg/L, and <332 ng/L respectively. For stage I patients both cTnT or cTnI and NT-proBNP are below the threshold. For stage II patients either troponin or NT-proBNP are above the threshold.

Patients eligible for SCT with melphalan 200 mg/m2 who decline transplant will be considered an additional stratum and randomized separately.

Thus, there will be the following strata:

0.patients eligible for SCT with melphalan 200 mg/m2 who decline transplant,

1. cardiac stage I,
2. cardiac stage II.

After stratification, patients will then be randomized to receive either A: MDex:oral melphalan at 0.22 mg/kg and dexamethasone at 40 mg daily for 4 consecutive days every 28 days (MDex) or B: BMDex:cycles 1 and 2 = MDex with bortezomib at 1.3 mg/m2 i.v. on days 1, 4, 8 and 11 of a 28 day cycle,cycles 3 - 8 = MDex with bortezomib at 1.3 mg/m2 i.v. on days 1, 8, 15 and 22 of a 35 day cycle.

Treatment will start within 2 weeks after randomization.

Treatment is continued until

* completion of MDex cycle 9 or BMDex cycle 8 or
* achievement of a complete hematologic response after cycle 6 or
* achievement of a partial hematologic response and an organ response after cycle 6 or
* less than a partial hematologic response after cycle 3 or
* progression of clonal plasma cell disease.

On the first day of each new treatment cycle and before each bortezomib dose, the patient will be evaluated for possible toxicities that may have occurred after the previous dose(s). Toxicities are to be assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.0. Dose modifications or delays will be made based on the toxicity experienced during the previous cycle of therapy or newly encountered on Day 1 of a cycle. Dose reduction steps are presented.

The start of a new cycle can be delayed on a weekly basis (for a maximum of 3 weeks)until recovery from toxicity to a level allowing continuation of therapy. Delay of a new cycle for more than 3 weeks can only occur if a clear clinical benefit has been observed. Otherwise, if there is a delay in the start of a new cycle of more than 3 weeks due to insufficient recovery from toxicity, subjects will discontinue study drug and have procedures performed as outlined for the End of Treatment Visit in the Schedule of Events.

During treatment, prophylactic medications will include acyclovir 400 mg twice daily with dose adjusted for renal function, ciprofloxacin 250 mg twice a day on days 1-7 of each cycle, and a proton-pump inhibitor. Supportive measures will be used. Patients will be seen in clinic by their physicians prior to beginning each cycle of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of amyloidosis.
* Genetic testing must be negative for transthyretin mutations associated with hereditary amyloidosis or immunohistochemistry of amyloid deposits must provide clear evidence of kappa or lambda light chains in those who present with peripheral neuropathy or heart as the dominant organ involvement.
* Not eligible for ASCT with melphalan 200 mg/m2. Patients who are eligible for SCT with melphalan 200 mg/m2 but decline the procedure, can be enrolled in the study, but are stratified in a separate stratum before randomization.
* Patients must be 18 years of age.
* ECOG performance status 0,1 or 2.
* Measurable disease; al least one of the following criteria:
* monoclonal protein >10 g/L in serum,
* amyloid-forming (involved) FLC >75 mg/L with an abnormal K/L ratio,
* difference between involved and uninvolved FLC >50 mg/L,
* bone marrow with a clonal predominance.
* Symptomatic organ involvement (heart, kidney, liver/GI tract, peripheral nervous system). Definition of organ involvement is defined.
* Hemoglobin ≥11 g/dL, absolute neutrophil count ≥1500/mikroL, platelets ≥140,000/mikroL.
* Total bilirubin <2.5 mg/dL, alkaline phosphatase <5 × u.l.n., ALT <3 × u.l.n..
* Estimated glomerular filtration rate (eGFR) by the MDRD formula >30 ml/min.
* Only patients who are informed of the investigational nature of this study and sign and give written informed consent in accordance with institutional, national and European guidelines are eligible to participate.
* Women must be either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e. a hormonal contraceptive, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study. All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy.
* Men must agree to use an acceptable method for contraception for the duration of the study.

Exclusion Criteria:

* Amyloid-specific syndrome, such as carpal tunnel syndrome or skin purpura as the only evidence of disease. The finding of isolated vascular amyloid in a bone marrow biopsy specimen or in a plasmacytoma is not indicative of systemic amyloidosis.
* Isolated soft tissue involvement.
* Presence of non-AL amyloidosis.
* Previous treatment for plasma cell disease. A single previous cycle of dexamethasone or steroid equivalent (maximum cumulative dexamethasone dose 160 mg) is allowed; in this case baseline data must be obtained after steroid administration. Previous stem cell harvest is allowed, provided that mobilization is performed with G-CSF only.
* Bone marrow plasma cells >30%.
* Cardiac stage III disease: both cTnT > 0.035 ng/mL (or in place of cTnT the cTnI > 0.10 ng/mL) AND simultaneous NT-proBNP >332 ng/L. These subject can be enrolled in the ancillary phase II study.
* Repetitive ventricular arrhythmias on 24h Holter ECG in spite of anti-arrhythmic treatment.
* Chronic atrial fibrillation
* Supine systolic blood pressure <100 mmHg or symptomatic orthostatic hypotension or clinically important autonomic disease
* Grade 3 sensory or grade 1 painful peripheral neuropathy.
* Patients with AL who are eligible for ASCT with 200 mg/m2 of melphalan. These are patients <65 years of age, without cardiac involvement (determined according to the consensus criteria), with eGFR >51mL/min, left ventricular ejection fraction >45%, and bilirubin <2.0 mg/dL. Patients who are eligible for SCT with melphalan 200 mg/m2 but decline the procedure, can be enrolled in the study, but are stratified in a separate stratum before randomization.
* Pregnant or nursing women.
* Clinically overt multiple myeloma with lytic bone lesions
* Patients with uncontrolled infection or active malignancy with the exception of adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years.
* Patients with medically documented cardiac syncope, uncompensated NYHA Class 3 or 4 congestive heart failure, or myocardial infarction within the previous 6 months are not eligible.
* HIV positive.
* Patients with serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Patients with hypersensitivity to bortezomib, boron or mannitol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-01; Primary Completion 2016-02 (Actual); Study Completion 2016-07-31 (Actual)

PRIMARY OUTCOMES:
Number of Patients in CR and PR measured by level of serum light chain monoclonal protein | 3 cycles of therapy
  As defined by the International Society for Amyloidosis consensus.
  Complete response:
  * serum and urine IF negative,
  * normal FLC ratio,
  * bone marrow PC <5%
  Partial response if:
  * serum monoclonal >0.5 g/dL, a 50% reduction,
  * FLC in urine visible and >100 mg/day and 50% reduction,
  * FLC >2 times upper normal and 50% reduction.
  Progressive disease
  * from CR, abnormal FLC ratio
  * from PR or stable disease, 50% increase in monoclonal protein to >0.5 g/dL, or 50% increase in urine to >200 mg/day, or FLC increase of 50% to >100 mg/L.
  Stable disease: no CR, no PR, no progression.

SECONDARY OUTCOMES:
Compare haematology response | 2 years
  To compare in patients treated with MDex or BMDex:
  * complete hematologic response rate after 3 cycles and after completion of therapy;
  * hematologic response rate at completion of therapy;
  * organ response rates at 3, 6, 9 and 12 months;
  * treatment-related mortality;
  * toxicity;
  * overall and progression-free survival;
  * time to hematologic and organ response;
  * quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni mr Palladini, Proff, Principal Investigator — Amyloidosis Research and Treatment Center, Pavia, Italy
Locations (1):
- Amyloidosis Research and Treatment Center, Pavia, Italy

REFERENCES:
- [Result] Kastritis E, Wechalekar AD, Dimopoulos MA, Merlini G, Hawkins PN, Perfetti V, Gillmore JD, Palladini G. Bortezomib with or without dexamethasone in primary systemic (light chain) amyloidosis. J Clin Oncol. 2010 Feb 20;28(6):1031-7. doi: 10.1200/JCO.2009.23.8220. Epub 2010 Jan 19. PMID 20085941
- [Derived] Kastritis E, Leleu X, Arnulf B, Zamagni E, Cibeira MT, Kwok F, Mollee P, Hajek R, Moreau P, Jaccard A, Schonland SO, Filshie R, Nicolas-Virelizier E, Augustson B, Mateos MV, Wechalekar A, Hachulla E, Milani P, Dimopoulos MA, Fermand JP, Foli A, Gavriatopoulou M, Klersy C, Palumbo A, Sonneveld P, Johnsen HE, Merlini G, Palladini G. Bortezomib, Melphalan, and Dexamethasone for Light-Chain Amyloidosis. J Clin Oncol. 2020 Oct 1;38(28):3252-3260. doi: 10.1200/JCO.20.01285. Epub 2020 Jul 30. PMID 32730181
- See also: "Click here for more information about this study:" EMN-03 — http://www.myeloma-europe.org/